CLINICAL TRIAL: NCT04610671
Title: A Phase 1 Study of CG0070 Combined With Nivolumab in Cisplatin Ineligible Patients With Muscle Invasive Bladder Cancer (MIBC)
Brief Title: Study of CG0070 Combined With Nivolumab in Cisplatin Ineligible Patients With MIBC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: CG Oncology, Inc. (Industry); Richard M. Shulze Family Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20575
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Muscle-Invasive Bladder Carcinoma; Bladder Cancer
Keywords: Bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants Receiving CG0070 & Nivolumab (Experimental): Both CG0070 (x 6 instillations) and nivolumab (x 2 doses) will be administered at their single-agent dose and schedule.
  Interventions: Drug: CG0070; Drug: Nivolumab

INTERVENTIONS:
Drug: CG0070 — CG0070 will be administered at a dose of 1x10^12 vp intravesically following a sequence of bladder washes with 5% DDM and normal saline.
Drug: Nivolumab — Two neoadjuvant doses of nivolumab 480 mg Q4W (every 4 weeks) for 2 doses (week 2 and 6)

SUMMARY:
Investigators will evaluate the safety and efficacy of combination neoadjuvant therapy using intravesical CG0070 and IV Nivolumab in cisplatin ineligible patients with Muscle Invasive Bladder Cancer (MIBC).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed MIBC (T2-T4a, N0-N1, M0 per American Joint Commission on Cancer [AJCC]) pure or mixed histology urothelial carcinoma. Clinical node- positive (N1) patients are eligible provided the lymph nodes (LNs) are within the planned surgical LN dissection template.
* The initial TURBT that showed muscularis propria invasion should be within 90 days prior to beginning study therapy. Participants must have sufficient baseline tumor tissue from either initial or repeat TURBTs. The local site pathologist will be asked to estimate and record the rough approximate percentage of viable tumor in the TURBT sample (initial or repeat TURBT with highest tumor content) to document at least 20% viable tumor content prior to registration. This is to ensure adequate tissue is available to perform tumor infiltrating CD8+ T-cell assessment. (The actual CD8+ T cell analysis will be done by a Central Laboratory and will not be done prior to registration.)
* Participants must be ineligible for cisplatin-based chemotherapy due to any of the following:

  * Creatinine clearance (CrCl) < 60 mL/min (with ECOG Performance Status (PS) 0-1)
  * Hearing impaired ≥ Grade 2 by CTCAE criteria
  * Neuropathy ≥ Grade 2 by CTCAE criteria
  * Heart failure NYHA ≥ III
  * ECOG ≥ 2
  * Refusing to undergo cisplatin chemotherapy
* Participants must be medically fit for TURBT and radical cystectomy (RC)
* Age ≥ 18 years
* Ability to understand and willingness to sign IRB-approved informed consent
* Willing to provide tumor tissue, blood, and urine samples for research
* Adequate organ function as measured by the following criteria, obtained ≤ 4 weeks prior to registration:

  * Absolute Neutrophil Count (ANC) ≥ 1000/mm3 (stable off growth factor within 4 weeks of first study drug administration)
  * Platelets ≥ 100,000/mm3
  * Hemoglobin ≥ 8 g/dL
  * Serum Creatinine Clearance ≥ 20 mL/min using the Cockcroft-Gault formula
  * ALT and AST ≤ 2.5x ULN
  * Total Bilirubin ≤ 1.5x ULN (in the absence of previously diagnosed Gilbert's disease)

Exclusion Criteria:

* Women who are pregnant or breastfeeding, since the effects of nivolumab and CG0070 on the fetus or breastfeeding child are unknown. All sexually active females of childbearing potential (not surgically sterilized and between menarche and 1 year post menopause) must have a blood test to rule out pregnancy within 4 weeks prior to registration.
* Participant with local symptoms from bladder cancer, (e.g. gross hematuria, dysuria, etc.) who are deemed to be unable to complete the treatment protocol.
* Participant with active or prior documented autoimmune disease within the past 2 years prior to Screening or other immunosuppressive agent within 14 days of study treatment. NOTE: Participant with well controlled type 1 diabetes mellitus, vitiligo, Graves disease, Hashimoto's disease, eczema, lichen simplex chronicus, or psoriasis not requiring systemic treatment (within the past 2 years prior to Screening) are not excluded
* Participants who have concurrent upper urinary tract (i.e. ureter, renal pelvis) invasive urothelial carcinoma. Participants with history of non-invasive (Ta, T1, Tis) upper tract urothelial carcinoma that has been definitively treated with at least one post-treatment disease assessment (i.e. cytology, biopsy, imaging) that demonstrates no evidence of residual disease are eligible.
* Participants who have another malignancy that could interfere with the evaluation of safety or efficacy of the study drugs. Participants with a prior malignancy will be allowed without Principle Investigator approval in the following circumstances:

  * Not currently active and diagnosed at least 3 years prior to the date of registration.
  * Non-invasive diseases such as low risk cervical cancer or any cancer in situ.
  * Localized (early stage) cancer treated with curative intent (without evidence of recurrence and intent for further therapy), and in which no chemotherapy was indicated (e.g. low/intermediate risk prostate cancer, etc.). Participants with other malignancies not meeting these criteria must be discussed prior to registration.
* Participants who have received any prior immune checkpoint inhibitor (i.e. anti-KIR, anti-PD-1, anti- PD-L1, anti-CTLA4 or other).
* Participants who have undergone major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury or specific anti-cancer treatment ≤ 4 weeks prior to starting study drug, or patients who have had placement of vascular access device ≤ 1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury.
* Participants who have clinically significant cardiac diseases deemed not fit for radical cystectomy, including any of the following:

  * History or presence of serious uncontrolled ventricular arrhythmias.
  * Clinically significant resting bradycardia.
  * Any of the following within 3 months prior to starting study drug: severe/unstable angina, Congestive Heart Failure (CHF), Cerebrovascular Accident (CVA), Transient Ischemic Attack (TIA).
  * Uncontrolled hypertension defined by a SBP ≥ 180 mm Hg and/or DBP ≥ 100 mm Hg, with or without anti-hypertensive medication(s).
* Participants who have history of chronic active liver disease or evidence of acute or chronic Hepatitis B Virus (HBV) or Hepatitis C (HCV).
* Participants who have known diagnosis of human immunodeficiency virus (HIV) infection. Testing is not required in absence of clinical suspicion.
* Participants who have known diagnosis of any condition (e.g. post-hematopoietic or solid organ transplant, pneumonitis, inflammatory bowel disease, etc.) that requires chronic immunosuppressive therapy which cannot be stopped for the duration of the clinical trial. Usage of non-steroidal anti-inflammatory medications (NSAIDS) for the treatment of osteoarthritis and uric acid synthesis inhibitors for the treatment of gout are permitted.
* Participants with any serious and/or uncontrolled concurrent medical conditions (e.g. active or uncontrolled infection, uncontrolled diabetes) or psychiatric illness that could, in the investigator's opinion, cause unacceptable safety risks or potentially interfere with the completion of the treatment according to the protocol.
* Participants who have used any live viral vaccine for prevention of infectious diseases within 4 weeks prior to study drug(s). Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, BCG, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
* Participants unwilling or unable to comply with the protocol.
* Participants with a known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Participants who participate in any other therapeutic clinical trials, including those with other investigational agents not included in this trial throughout the duration of this study.
* Use of excluded antiviral medication that cannot be suspended at least 14 days prior and for 14 days after the administration of any CG0070 treatment throughout the duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2025-01-18 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Up to 24 months after start of treatment
  Adverse events Grade 3 or higher will be graded according to the NC Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0

SECONDARY OUTCOMES:
Change in PD-L1 expression on tumor and immune cells | Up to 24 months after start of treatment
  The change in PD-L1 expression on tumor and immune cells from pre-treatment TURBT to post- treatment cystectomy samples will be assessed and analyzed using McNemar test for the change in the percentage of PD-L1 positivity before and after the study treatment, using the Stuart-Maxwell test with 4 ordered categories.

OTHER OUTCOMES:
Changes in intraepithelial CD8+ T cell density | Up to 24 months after start of treatment
  The changes in intraepithelial CD8+ T cell density from pre-treatment TURBT to post-treatment cystectomy samples will be assessed using a paired t-test or Wilcoxon signed rank test according to the distribution of changes in the CD8+T cell density. The distribution of changes will be investigated using the Anderson-Darling test.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Li, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- [Result] Li R, Villa NY, Yu X, Johnson JO, Borjas G, Dhillon J, Moran-Segura CM, Kim Y, Francis N, Dorman D, Powers JJ, Sexton WJ, Spiess PE, Poch MA, Zemp L, Gilbert SM, Zhang J, Pow-Sang JM, Anderson ARA, Li T, Wang X, Grass GD, Burke JM, Dinney CPN, Rodriguez PC, Jain RK, Mule JJ, Conejo-Garcia JR. Oncolytic immunotherapy with nivolumab in muscle-invasive bladder cancer: a phase 1b trial. Nat Med. 2025 Jan;31(1):176-188. doi: 10.1038/s41591-024-03324-9. Epub 2024 Nov 9. PMID 39521884

DOCUMENTS (1):
  • Informed Consent Form (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT04610671/ICF_000.pdf